CLINICAL TRIAL: NCT01083225
Title: Randomised Controlled Trial on the Effect of Individual User Involvement in a Mental Health Center
Brief Title: Effect of Patient Participation in Mental Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other); The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008/2/0325
Record Dates: First submitted 2010-02-23; First posted 2010-03-09 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Client feedback (Experimental)
  Interventions: Behavioral: Client feedback
- Treatment as usual (Active Comparator)
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Client feedback — Client feedback during consultations using ORS (Outcome rating scale) and SRS (Session rating scale).
  Arms: Client feedback
Behavioral: Treatment as usual — Treatment as usual, consultations
  Arms: Treatment as usual

SUMMARY:
The purpose of this study is to evaluate the effect of individual user involvement in an outpatient mental health center. The intervention consists of patients completing a self-report symptom and problem questionnaire and reviewing it with a clinician.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.

Exclusion Criteria:

* Not able to complete the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Mental health symptom score (Basis-32) | Baseline, 6 weeks, 6 months & 12 months
Patient activation (Patient Activation Measure) | Baseline, 6 weeks, 6 months & 12 months
Alliance (Inpatient treatment alliance scale) | Baseline, 6 weeks, 6 months & 12 months

SECONDARY OUTCOMES:
Patient satisfaction (Client Satisfaction Questionnaire) | Baseline, 6 weeks, 6 months & 12 months
Quality of life (Short form 12) | Baseline, 6 weeks, 6 months & 12 months
Evaluation of problems (Outcome rating scale) | Baseline, 6 weeks, 6 months & 12 months
Evaluation of consultations (Session Rating Scale) | Baseline, 6 weeks, 6 months & 12 months
Evaluation of involvement | Baseline, 6 weeks, 6 months & 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Aslak Steinsbekk, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St. Olavs Hospital, Nidaros Mental Health Center, Trondheim, Norway

REFERENCES:
- [Result] Rise MB, Eriksen L, Grimstad H, Steinsbekk A. The long-term effect on mental health symptoms and patient activation of using patient feedback scales in mental health out-patient treatment. A randomised controlled trial. Patient Educ Couns. 2016 Jan;99(1):164-8. doi: 10.1016/j.pec.2015.07.016. Epub 2015 Jul 19. PMID 26227577